CLINICAL TRIAL: NCT01852656
Title: The Effectiveness and Cost of Different Methods of Reminders for Annual Influenza Immunization Among Adults With Asthma and Chronic Obstructive Pulmonary Disease
Brief Title: Effectiveness of Influenza Vaccine Reminder Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12010936
Record Dates: First submitted 2012-10-08; First posted 2013-05-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: Influenza, Human; Immunization
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Postcard Only Reminder Group (Active Comparator): In the postcard reminder intervention, the member will receive a single postcard, addressed to the member with asthma or COPD.
  Interventions: Behavioral: Postcard Only Reminder Group
- IVR Only Reminder Group (Active Comparator): In the IVR reminder intervention, targeted members will be contacted by the interactive voice response system
  Interventions: Behavioral: IVR Only Reminder Group
- Postcard and IVR Reminder Group (Active Comparator): In this group, individuals will receive both a postcard reminder and an IVR reminder.
  Interventions: Behavioral: Postcard and IVR Reminder Group

INTERVENTIONS:
Behavioral: Postcard and IVR Reminder Group — IVR: Subjects in this reminder group will receive an automated telephone call to their primary telephone number. A total of 2 call attempts per member will be made. The IVR system will provide a message about the importance of annual influenza vaccination. The member can also request additional information about influenza vaccination and influenza vaccination locations and times.
  Postcard: The postcard will be sent as a single postcard to each individual on the list. The postcard will be sent to the home address of the member. If the postcard is returned, the postcard will not be re-sent. The postcard does not identify that the member has a chronic health condition such as asthma or COPD. The postcard will be mailed during the last two weeks of September, 2012.
  Arms: Postcard and IVR Reminder Group
Behavioral: Postcard Only Reminder Group — Postcard: The postcard will be sent as a single postcard to each individual on the list. The postcard will be sent to the home address of the member. If the postcard is returned, due to an inaccurate address, the postcard will not be re-sent. The postcard does not identify that the member has a chronic health condition such as asthma or COPD. The postcard will be mailed during the last two weeks of September, 2012.
  Arms: Postcard Only Reminder Group
Behavioral: IVR Only Reminder Group — IVR: Subjects in this reminder group will receive an automated telephone call to their primary telephone number. A total of 2 call attempts per member will be made. The IVR system will provide a message about the importance of annual influenza vaccination. The member can also request additional information about influenza vaccination and influenza vaccination locations and times.
  Arms: IVR Only Reminder Group

SUMMARY:
Influenza disease causes significant morbidity and mortality in the Unites States each year. Although influenza can cause morbidity in otherwise healthy individuals, adults with chronic lung disease have significantly increased rates of hospitalization from influenza-related illnesses compared to healthy adults. Influenza vaccination is the primary means of preventing influenza disease. Annual influenza vaccination is recommended for all individuals 6 months of age and older in the United States. Influenza vaccination rates are sub-optimal, however. Patient reminder/recall has been shown, in multiple studies across a variety of age groups and health conditions, to increase immunization rates. However, the effectiveness and cost-effectiveness of different types of reminder/recall has not been well-studied, particularly in adults. In the fall of 2012, the Population and Prevention Services (PPS) Department at Kaiser Permanente Colorado (KPCO) is using 3 different reminder strategies for influenza vaccination among adults with asthma and chronic obstructive pulmonary disease (COPD). The objective of this study is to provide a rigorous evaluation of which strategy is more effective and more cost-effective, to promote influenza vaccination.

DETAILED DESCRIPTION:
At KPCO, postcards are typically sent to members each fall, to remind members to receive their annual influenza vaccine. At KPCO, interactive voice response (IVR) systems have been utilized for a number of prevention reminders, but have not in the past been used for influenza vaccination reminders. For the 2012-2013 influenza season, the PPS department is going to send three different types of reminders to their adult patients with certain chronic lung diseases (specifically, adults with asthma and COPD): postcards only; IVR reminders only; postcards plus IVR reminders. This study seeks to evaluate the effectiveness, and cost-effectiveness, of an already-finalized operational plan for influenza reminders.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 to 64 years
* Enrolled in Kaiser Permanente Colorado health plan
* Diagnosis of asthma and/or chronic obstructive pulmonary disease

Exclusion Criteria:

* Subjects living in households with other individuals in high-risk categories for influenza morbidity

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12255 (Actual)
Dates: Start 2012-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Receipt of influenza vaccine | up to 7 months
  The 2012-2013 influenza season, defined as October to April.

SECONDARY OUTCOMES:
Total unit cost per outreach method | up to 10 months
  The time in months to develop, plan, and implement the intervention arms, as a function of cost.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew F. Daley, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Colorado, Denver, Colorado, United States